CLINICAL TRIAL: NCT01937156
Title: A Randomized, Active-control, Double-blind, Double-dummy, Parallel-group, Multi-center Study to Assess the Efficacy and Safety of SP-01 (Granisetron Transdermal Delivery System) in Chemotherapy-induced Nausea and Vomiting Associated With the Administration of Moderately or Highly Emetogenic (ME or HE) Multi-day Chemotherapy
Brief Title: A Randomized Controlled Trial of SP-01 (Granisetron Transdermal Delivery System) in Chemotherapy-induced Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solasia Pharma K.K. (Industry)
Collaborators: Proswell Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SP-0103
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Granisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP-01 (Experimental)
  Interventions: Drug: SP-01 (Granisetron Transdermal Delivery System)
- Granisetron Hydrochloride Tablet (Active Comparator)
  Interventions: Drug: Granisetron Hydrochloride Tablet

INTERVENTIONS:
Drug: SP-01 (Granisetron Transdermal Delivery System) — SP-01 will be applied to the upper arm 24-48 hours before the start of chemotherapy, and left in place for 7 days.
  Arms: SP-01
Drug: Granisetron Hydrochloride Tablet — Granisetron hydrochloride 1 mg tablets will be administered 1 hour before administration of chemotherapy at the first time, then taken 12 hours after the first dose later; 2 mg/day bid, for ≥ 2 days.
  Arms: Granisetron Hydrochloride Tablet

SUMMARY:
The purpose of this study is to assess the efficacy and safety of SP-01 in chemotherapy-induced nausea and vomiting (CINV) associated with the administration of moderately or highly emetogenic (ME or HE) multi-day chemotherapy，which will provide scientific and reliable clinical data in the drug registration in China.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18years
* Histologically and/or cytologically confirmed cancer
* The physical status score ECOG ≤ 2
* Life expectancy of ≥3 months
* Will receive multi-day ME/HE chemotherapy (≥2 days) with the emetogenic potential of level 3-5
* In accordance with the indication of chemotherapy and basic requirements;

  * Peripheral Haematology: Hb ≥ 9.0 g/dL, absolute neutrophil count ≥ 1.5×10e9/L, platelet count ≥ 80×10e9/L
  * Blood biochemistry: Total bilirubin < 1.25×ULN, ALT and AST ≤ 2.5×ULN; if liver metastasis, ALT and AST < 5×ULN, Creatinine ≤ 1×ULN, basic normal serum electrolyte (Na, Ka, Cl, Ca)
  * Other important organs function normally
* Subjects voluntarily participate and signed the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving Complete Control (CC) of CINV from the first administration until 24 hour after the last administration of ME or HE multi-day chemotherapy | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, MD, Principal Investigator — The 81st hospital of P.L.A.
Locations (1):
- The 81st Hospital of P.L.A., Nanjing, Jiangsu, China